CLINICAL TRIAL: NCT04084613
Title: Mepolizumab: Real World Evidence Study for the Treatment of Severe Eosinophilic Asthma in Greece
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Stylianos Loukides, Assistant Professor, Attikon Hospital
Other Study IDs: Mepolizumab RWE Study Greece
Record Dates: First submitted 2019-09-08; First posted 2019-09-10 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Severe Eosinophilic Asthma
Keywords: Severe Eosinophilic Asthma; Mepolizumab; Anti-IL5 treatment
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with uncontrolled severe eosinophilic asthma: Asthmatic patients with peripheral blood eosinophils ≥300 cells/μL at any measurement in the previous year or ≥150 cells/μL in a recent measurement, with poor symptom control and increased number of exacerbations (2 or more) despite optimal treatment with high doses of inhaled corticosteroids and β2 stimulants.

SUMMARY:
A prospective multi-centre, non-interventional observational study, that will be conducted in several centers in Greece for a 2-year time period (completion date December 2020), to describe patient characteristics, medical history, and the clinical benefit of mepolizumab in patients with severe eosinophilic asthma newly initiated to the drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncontrolled severe eosinophilic asthma placed under treatment with mepolizumab, i.e. in patients with peripheral blood eosinophils ≥300 cells/μL at any measurement in the previous year or ≥150 cells/μL in a recent measurement, with poor symptom control and increased number of exacerbations (2 or more) despite optimal treatment with high doses of inhaled corticosteroids and β2 stimulants

Exclusion Criteria:

* Patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with uncontrolled severe eosinophilic asthma
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of annual exacerbation rate in patients with severe eosinophilic asthma in treatment with mepolizumab | 2 years
  Reduction of the clinical significant exacerbations in comparison to the year before the initiation of treatment with mepolizumab. A clinical significant exacerbation is an exacerbation that requires treatment as follows: increase of dose of oral corticosteroids intake
Quality of life improvement in patients with severe eosinophilic asthma receiving mepolizumab as it measured by Asthma Control Test (ACT) | 2 years
  ACT is a 5-point scale that assesses the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control. An ACT score 19 or less means that asthma is not well controlled

IPD SHARING:
Plan to Share IPD: No